CLINICAL TRIAL: NCT01766206
Title: A Multicenter Post Marketing Surveillance Study to Monitor the Safety of GlaxoSmithKline (GSK) Biologicals' Meningococcal ACWY Conjugate Vaccine(MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects From 2 Months to 55 Years of Age in the Republic of South Korea.
Brief Title: Safety of One Dose of Meningococcal ACWY Conjugate Vaccine in Subjects From 2 Months to 55 Years of Age in the Republic of South Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205341; V59_62 (Other: Novartis)
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-07

CONDITIONS: Meningococcal Disease
Keywords: conjugate vaccine; phase IV clinical trial; Neisseria meningitidis
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- MenACWY-CRM Group (Experimental): Healthy subjects from 2 months to 55 years of age in South Korea, who received MenACWY-CRM (Menveo) vaccination, according to routine clinical care.
  Interventions: Biological: MenACWY-CRM (Menveo)

INTERVENTIONS:
Biological: MenACWY-CRM (Menveo) — One dose administered intramuscularly preferably into the anterolateral aspect of the thigh in infants or into the deltoid muscle in children, adolescents and adults.

SUMMARY:
A multicenter, single arm, post-marketing surveillance study. This study is a postlicensure requirement of the Korea Food and Drug Administration (KFDA) to provide continued safety evaluation of MenACWY in the Korean population from 2 months to 55 years of age, receiving MenACWY-CRM vaccination according to routine clinical practice and prescribing information.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrolment in this study are those:

1. male and female subjects from 2 months to 55 years of the age at the time of Visit 1 (including all 55 years old subjects, up to one day before their 56th year birthday), who are scheduled to receive vaccination with MenACWY-CRM conjugate vaccine, according to the local prescribing information and routine clinical practice;
2. to whom the nature of the study has been described and the subject or subject's parent/legal representative has provided written informed consent;
3. whom the investigator believes that the subject can and will comply with the requirements of the protocol (e.g., completion of the Diary Card);
4. who are in good health as determined by the outcome of medical history, physical assessment and clinical judgment of the investigator.

Exclusion Criteria:

1. Contraindication, special warnings and/or precautions, as evaluated by the investigators, reported in the MenACWY-CRM conjugate vaccine Korean prescribing information. In particular, should not be included in the study a subject who has ever had:

* an allergic reaction to the active substances or any of the other ingredients of the study vaccine; an allergic reaction to diphtheria toxoid;
* an illness with high fever; however, a mild fever or upper respiratory infection (for example cold) itself is not a reason to delay vaccination. Special care should be taken for subjects having haemophilia or any other problem that may stop your blood from clotting properly, such as persons receiving blood thinners (anticoagulants).

Ages: 2 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3948 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- South Korea (22):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Anyang
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Changwon
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Donghae
  - GSK Investigational Site, Gimhae
  - GSK Investigational Site, Goyang-si
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Guro Gu
  - GSK Investigational Site, Gwangmyeong
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeju City
  - GSK Investigational Site, Jeollanam Do
  - GSK Investigational Site, Kyeonggido
  - GSK Investigational Site, Pyeongtaek-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
  - GSK Investigational Site, Yangju-si, Gyeonggi-do

REFERENCES:
- [Background] Al-Tawfiq JA, Clark TA, Memish ZA. Meningococcal disease: the organism, clinical presentation, and worldwide epidemiology. J Travel Med. 2010 Sep-Oct;17 Suppl:3-8. doi: 10.1111/j.1708-8305.2010.00448.x. No abstract available. PMID 20849427
- [Background] Bae SM, Kang YH. Serological and genetic characterization of meningococcal isolates in Korea. Jpn J Infect Dis. 2008 Nov;61(6):434-7. PMID 19050348
- [Background] Cho HK, Lee H, Kang JH, Kim KN, Kim DS, Kim YK, Kim JS, Kim JH, Kim CH, Kim HM, Park SE, Oh SH, Chung EH, Cha SH, Choi YY, Hur JK, Hong YJ, Lee HJ, Kim KH. The causative organisms of bacterial meningitis in Korean children in 1996-2005. J Korean Med Sci. 2010 Jun;25(6):895-9. doi: 10.3346/jkms.2010.25.6.895. Epub 2010 May 24. PMID 20514311
- [Background] Deasy A, Read RC. Challenges for development of meningococcal vaccines in infants and children. Expert Rev Vaccines. 2011 Mar;10(3):335-43. doi: 10.1586/erv.11.3. PMID 21434801
- [Background] Hill DJ, Griffiths NJ, Borodina E, Virji M. Cellular and molecular biology of Neisseria meningitidis colonization and invasive disease. Clin Sci (Lond). 2010 Feb 9;118(9):547-64. doi: 10.1042/CS20090513. PMID 20132098
- [Background] Lee JH, Cho HK, Kim KH, Kim CH, Kim DS, Kim KN, Cha SH, Oh SH, Hur JK, Kang JH, Kim JH, Kim YK, Hong YJ, Chung EH, Park SE, Choi YY, Kim JS, Kim HM, Choi EH, Lee HJ. Etiology of invasive bacterial infections in immunocompetent children in Korea (1996-2005): a retrospective multicenter study. J Korean Med Sci. 2011 Feb;26(2):174-83. doi: 10.3346/jkms.2011.26.2.174. Epub 2011 Jan 24. PMID 21286006
- [Background] Moon SY, Chung DR, Kim SW, Chang HH, Lee H, Jung DS, Kim YS, Jung SI, Ryu SY, Heo ST, Moon C, Ki HK, Son JS, Kwon KT, Shin SY, Lee JS, Lee SS, Rhee JY, Lee JA, Joung MK, Cheong HS, Peck KR, Song JH. Changing etiology of community-acquired bacterial meningitis in adults: a nationwide multicenter study in Korea. Eur J Clin Microbiol Infect Dis. 2010 Jul;29(7):793-800. doi: 10.1007/s10096-010-0929-8. Epub 2010 May 1. PMID 20432052
- [Background] Obaro SK, Madhi SA. Bacterial pneumonia vaccines and childhood pneumonia: are we winning, refining, or redefining? Lancet Infect Dis. 2006 Mar;6(3):150-61. doi: 10.1016/S1473-3099(06)70411-X. PMID 16500596
- [Background] Rouphael NG, Stephens DS. Neisseria meningitidis: biology, microbiology, and epidemiology. Methods Mol Biol. 2012;799:1-20. doi: 10.1007/978-1-61779-346-2_1. PMID 21993636
- [Background] Trotter CL, Andrews NJ, Kaczmarski EB, Miller E, Ramsay ME. Effectiveness of meningococcal serogroup C conjugate vaccine 4 years after introduction. Lancet. 2004 Jul 24-30;364(9431):365-7. doi: 10.1016/S0140-6736(04)16725-1. PMID 15276396
- [Derived] Yoo BW, Jung HL, Byeon YS, Han DK, Jeong NY, Curina C, Moraschini L, Kim SJ, Bhusal C, Pellegrini M, Miao Y. Results from a large post-marketing safety surveillance study in the Republic of Korea with a quadrivalent meningococcal CRM-conjugate vaccine in individuals aged 2 months-55 years. Hum Vaccin Immunother. 2020 Jun 2;16(6):1260-1267. doi: 10.1080/21645515.2019.1670125. Epub 2019 Oct 25. PMID 31634044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects from 2 months to 55 years of age were enrolled in 46 centres in South Korea.
Pre-assignment Details: Out of the 3,948 subjects enrolled, only 3,939 subjects were exposed to vaccination as 1 subject did not receive a study vaccination and 8 subjects did not provide post vaccination safety data. Among 3939 subjects, 15 subjects are in the ≥ 56 age category (outside the range defined as per the protocol).
Period: Overall Study
Arm/Group | MenACWY-CRM Group
Started (Among 3939 subjects, 15 are in the ≥ 56 age category (outside the range defined as per the protocol)) | 3939
Completed | 3888
Not Completed | 51
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 10
Not completed — Inappropriate enrollment | 18
Not completed — Withdrawal and inappropriate enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | MenACWY-CRM Group
Number analyzed (Participants) | 3939
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.37 (15.4)
Age, Customized [Number; unit: Participants]
  2- 23 months | 654
  2-10 years | 890
  2-5 years | 551
  6-10 years | 339
  11-18 years | 433
  19-34 years | 1286
  35 - 55 years | 661
  ≥ 56 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2181
  Male | 1758
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3937
  Caucasian | 1
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Local and Systemic Solicited Adverse Events (AEs)
Description: Assessed solicited local AEs include: injection site erythema, injection site induration, injection site tenderness, injection site pain. Assessed solicited systemic AEs include: change in eating habits, sleepiness, irritability, rash, vomiting, diarrhea, fever, chills, nausea, malaise, generalized myalgia, generalized arthralgia, headache. "Any" is defined as any report of the specified symptom irrespective of intensity grade. Subjects from 2 months to 55 years of age were evaluated for the outcome measure.
Time Frame: From Day 1 of vaccination to Day 7 post vaccination
Population: This analysis was performed on the Safety per protocol set, which included enrolled subjects aged from 2 months to 55 years, who signed an informed consent, underwent screening, received a subject number and received a study vaccination and provided post vaccination data. Excluding 19 subjects from safety set with protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY-CRM Group
Number analyzed (Participants) | 3920
Participants
  Any injection site tenderness, 2 - 23 months: number analyzed (Participants) | 653
  Any injection site tenderness, 2 - 23 months | 67
  Any injection site erythema, 2 - 23 months: number analyzed (Participants) | 653
  Any injection site erythema, 2 - 23 months | 32
  Any injection site induration, 2 - 23 months: number analyzed (Participants) | 653
  Any injection site induration, 2 - 23 months | 28
  Any change in eating habbits, 2 - 23 months: number analyzed (Participants) | 653
  Any change in eating habbits, 2 - 23 months | 110
  Any sleepiness, 2 - 23 months: number analyzed (Participants) | 653
  Any sleepiness, 2 - 23 months | 126
  Any irritability, 2 - 23 months: number analyzed (Participants) | 653
  Any irritability, 2 - 23 months | 219
  Any vomiting, 2 - 23 months: number analyzed (Participants) | 653
  Any vomiting, 2 - 23 months | 66
  Any diarrhea, 2 - 23 months: number analyzed (Participants) | 653
  Any diarrhea, 2 - 23 months | 82
  Any rash, 2 - 23 months: number analyzed (Participants) | 653
  Any rash, 2 - 23 months | 20
  Any fever, 2 - 23 months: number analyzed (Participants) | 653
  Any fever, 2 - 23 months | 57
  Any injection site tenderness, 2 - 5 years: number analyzed (Participants) | 551
  Any injection site tenderness, 2 - 5 years | 135
  Any injection site erythema, 2 - 5 years: number analyzed (Participants) | 551
  Any injection site erythema, 2 - 5 years | 71
  Any injection site induration, 2 - 5 years: number analyzed (Participants) | 551
  Any injection site induration, 2 - 5 years | 49
  Any change in eating habits, 2 - 5 years: number analyzed (Participants) | 551
  Any change in eating habits, 2 - 5 years | 22
  Any sleepiness, 2 - 5 years: number analyzed (Participants) | 551
  Any sleepiness, 2 - 5 years | 17
  Any irritability, 2 - 5 years: number analyzed (Participants) | 551
  Any irritability, 2 - 5 years | 35
  Any vomiting, 2 - 5 years: number analyzed (Participants) | 551
  Any vomiting, 2 - 5 years | 4
  Any diarrhea, 2 - 5 years: number analyzed (Participants) | 551
  Any diarrhea, 2 - 5 years | 7
  Any rash, 2 - 5 years: number analyzed (Participants) | 551
  Any rash, 2 - 5 years | 18
  Any fever, 2 - 5 years: number analyzed (Participants) | 551
  Any fever, 2 - 5 years | 12
  Any injection site tenderness, 6 - 10 years: number analyzed (Participants) | 338
  Any injection site tenderness, 6 - 10 years | 108
  Any injection site erythema, 6 - 10 years: number analyzed (Participants) | 338
  Any injection site erythema, 6 - 10 years | 53
  Any injection site induration, 6 - 10 years: number analyzed (Participants) | 338
  Any injection site induration, 6 - 10 years | 45
  Any chills, 6 - 10 years: number analyzed (Participants) | 338
  Any chills, 6 - 10 years | 7
  Any nausea, 6 - 10 years: number analyzed (Participants) | 338
  Any nausea, 6 - 10 years | 7
  Any malaise, 6 - 10 years: number analyzed (Participants) | 338
  Any malaise, 6 - 10 years | 5
  Any myalgia, 6 - 10 years: number analyzed (Participants) | 338
  Any myalgia, 6 - 10 years | 6
  Any arthralgia, 6 - 10 years: number analyzed (Participants) | 338
  Any arthralgia, 6 - 10 years | 6
  Any headache, 6 - 10 years: number analyzed (Participants) | 338
  Any headache, 6 - 10 years | 11
  Any rash, 6 - 10 years: number analyzed (Participants) | 338
  Any rash, 6 - 10 years | 10
  Any fever, 6 - 10 years: number analyzed (Participants) | 338
  Any fever, 6 - 10 years | 9
  Any injection site tenderness, 11 - 18 years: number analyzed (Participants) | 431
  Any injection site tenderness, 11 - 18 years | 91
  Any injection site erythema, 11 - 18 years: number analyzed (Participants) | 431
  Any injection site erythema, 11 - 18 years | 17
  Any injection site induration, 11 - 18 years: number analyzed (Participants) | 431
  Any injection site induration, 11 - 18 years | 21
  Any chills, 11 - 18 years: number analyzed (Participants) | 431
  Any chills, 11 - 18 years | 9
  Any nausea, 11 - 18 years: number analyzed (Participants) | 431
  Any nausea, 11 - 18 years | 4
  Any malaise, 11 - 18 years: number analyzed (Participants) | 431
  Any malaise, 11 - 18 years | 9
  Any myalgia, 11 - 18 years: number analyzed (Participants) | 431
  Any myalgia, 11 - 18 years | 12
  Any arthralgia, 11 - 18 years: number analyzed (Participants) | 431
  Any arthralgia, 11 - 18 years | 5
  Any headache, 11 - 18 years: number analyzed (Participants) | 431
  Any headache, 11 - 18 years | 12
  Any rash, 11 - 18 years: number analyzed (Participants) | 431
  Any rash, 11 - 18 years | 6
  Any fever, 11 - 18 years: number analyzed (Participants) | 431
  Any fever, 11 - 18 years | 4
  Any injenction site tenderness, 19 - 34 years: number analyzed (Participants) | 1286
  Any injenction site tenderness, 19 - 34 years | 214
  Any injection site erythema, 19 - 34 years: number analyzed (Participants) | 1286
  Any injection site erythema, 19 - 34 years | 14
  Any injection site induration, 19 - 34 years: number analyzed (Participants) | 1286
  Any injection site induration, 19 - 34 years | 9
  Any chills, 19 - 34 years: number analyzed (Participants) | 1286
  Any chills, 19 - 34 years | 7
  Any nausea, 19 - 34 years: number analyzed (Participants) | 1286
  Any nausea, 19 - 34 years | 6
  Any malaise, 19 - 34 years: number analyzed (Participants) | 1286
  Any malaise, 19 - 34 years | 20
  Any myalgia, 19 - 34 years: number analyzed (Participants) | 1286
  Any myalgia, 19 - 34 years | 21
  Any arthralgia, 19 - 34 years: number analyzed (Participants) | 1286
  Any arthralgia, 19 - 34 years | 8
  Any headache, 19 - 34 years: number analyzed (Participants) | 1286
  Any headache, 19 - 34 years | 29
  Any rash, 19 - 34 years: number analyzed (Participants) | 1286
  Any rash, 19 - 34 years | 13
  Any fever, 19 - 34 years: number analyzed (Participants) | 1286
  Any fever, 19 - 34 years | 3
  Any injection site tenderness, 35 - 55 years: number analyzed (Participants) | 661
  Any injection site tenderness, 35 - 55 years | 174
  Any injection site erythema, 35 - 55 years: number analyzed (Participants) | 661
  Any injection site erythema, 35 - 55 years | 7
  Any injection site induration, 35 - 55 years: number analyzed (Participants) | 661
  Any injection site induration, 35 - 55 years | 6
  Any chills, 35 - 55 years: number analyzed (Participants) | 661
  Any chills, 35 - 55 years | 7
  Any nausea, 35 - 55 years: number analyzed (Participants) | 661
  Any nausea, 35 - 55 years | 9
  Any malaise, 35 - 55 years: number analyzed (Participants) | 661
  Any malaise, 35 - 55 years | 16
  Any myalgia, 35 - 55 years: number analyzed (Participants) | 661
  Any myalgia, 35 - 55 years | 23
  Any arthralgia, 35 - 55 years: number analyzed (Participants) | 661
  Any arthralgia, 35 - 55 years | 15
  Any headache, 35 - 55 years: number analyzed (Participants) | 661
  Any headache, 35 - 55 years | 19
  Any rash, 35 - 55 years: number analyzed (Participants) | 661
  Any rash, 35 - 55 years | 6
  Any fever, 35 - 55 years: number analyzed (Participants) | 661
  Any fever, 35 - 55 years | 2

2. Primary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment. All unsolicited AEs reported from day 1 to day 7 post vaccination were assessed. "Any" is defined as any report of the specified symptom irrespective of intensity grade. Subjects from 2 months to 55 years of age were evaluated for the outcome measure.
Time Frame: From Day 1 of vaccination to Day 7 post vaccination
Population: This analysis was performed on the Safety per protocol set, which included all enrolled subjects who signed an informed consent,underwent screening, received a subject number, received a study vaccination and provided post vaccination data. Excluding 19 subjects from safety set with protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY-CRM Group
Number analyzed (Participants) | 3920
Participants
  2 - 23 Months: number analyzed (Participants) | 653
  2 - 23 Months | 82
  2 - 5 Years: number analyzed (Participants) | 551
  2 - 5 Years | 56
  6 - 10 Years: number analyzed (Participants) | 338
  6 - 10 Years | 18
  11 - 18 Years: number analyzed (Participants) | 431
  11 - 18 Years | 8
  19 - 34 Years: number analyzed (Participants) | 1286
  19 - 34 Years | 17
  35 - 55 Years: number analyzed (Participants) | 661
  35 - 55 Years | 5

3. Primary Outcome: Number of Subjects Reporting Medically Attended AEs (MAAEs)
Description: MAAEs are defined as events that require a physician's visit or an emergency room visit. All reported MAAEs from day 1 to day 29 were assessed. Subjects from 2 months to 55 years of age were evaluated for the outcome measure.
Time Frame: From Day 1 of vaccination to study termination (Day 29/early termination)
Population: This analysis was performed on the Safety per protocol set, which included all enrolled subjects who signed an informed consent, underwent screening, received a subject number, received a study vaccination and provided post vaccination data. Excluding 19 subjects from safety set with protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY-CRM Group
Number analyzed (Participants) | 3920
Participants
  2 - 23 Months: number analyzed (Participants) | 653
  2 - 23 Months | 238
  2 - 5 Years: number analyzed (Participants) | 551
  2 - 5 Years | 120
  6 - 10 Years: number analyzed (Participants) | 338
  6 - 10 Years | 28
  11 - 18 Years: number analyzed (Participants) | 431
  11 - 18 Years | 20
  19 - 34 Years: number analyzed (Participants) | 1286
  19 - 34 Years | 16
  35 - 55 Years: number analyzed (Participants) | 661
  35 - 55 Years | 5

4. Primary Outcome: Number of Subjects Reporting Serious AEs (SAEs)
Description: An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening (i.e., the subject was, in the opinion of the investigator, at immediate risk of death from the event as it occurred); it does not refer to an event which hypothetically might have caused death if it were more severe, requires or prolongs subject's hospitalization, results in persistent or significant disability/incapacity (i.e., the event causes a substantial disruption of a person's ability to conduct normal life functions), results in a congenital anomaly/birth defect, is an important and significant medical event that may not be immediately life threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above. Subjects from 2 months to 55 years of age were evaluated for the outcome measure.
Time Frame: From Day 1 of vaccination to study termination (Day 29/early termination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY-CRM Group
Number analyzed (Participants) | 3920
Participants
  2 - 23 Months: number analyzed (Participants) | 653
  2 - 23 Months | 3
  2 - 5 Years: number analyzed (Participants) | 551
  2 - 5 Years | 3
  6 - 10 Years: number analyzed (Participants) | 338
  6 - 10 Years | 0
  11 - 18 Years: number analyzed (Participants) | 431
  11 - 18 Years | 2
  19 - 34 Years: number analyzed (Participants) | 1286
  19 - 34 Years | 0
  35 - 55 Years: number analyzed (Participants) | 661
  35 - 55 Years | 0

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs were reported from Day 1 to Day 7. MAAEs and SAEs were reported from study day 1 to study termination (Day 29/early termination).
Description: Total number of subjects at risk for SAEs, all cause mortality and FAEs were analyzed from the Safety set (including 15 subjects of ≥ 56 years age category).
Arm/Group | MenACWY-CRM Group
All-Cause Mortality (participants affected / at risk) | 0/3939
Serious Adverse Events (participants affected / at risk) | 8/3939
Other Adverse Events (participants affected / at risk) | 1379/3939
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM Group (N=3939)
Bronchiolitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM Group (N=3939)
Injection site tenderness (General disorders) | 202 (202) — This symptom was assessed as a solicited local AE.
Injection site pain (General disorders) | 592 (592) — This symptom was assessed as a solicited local AE.
Injection site erythema (General disorders) | 195 (195) — This symptom was assessed as a solicited local AE.
Injection site induration (General disorders) | 158 (158) — This symptom was assessed as a solicited local AE.
Eating disorder (Psychiatric disorders) | 132 (132) — This symptom was assessed as a solicited general AE.
Sleepiness (Nervous system disorders) | 143 (143) — This symptom was assessed as a solicited general AE.
Irritability (Psychiatric disorders) | 254 (254) — This symptom was assessed as a solicited general AE.
Vomiting (Gastrointestinal disorders) | 70 (70) — This symptom was assessed as a general AE.
Diarrhea (General disorders) | 89 (89) — This symptom was assessed as a solicited general AE.
Chills (General disorders) | 31 (31) — This symptom was assessed as a solicited general AE.
Nausea (General disorders) | 28 (28) — This symptom was assessed as a solicited general AE.
Malaise (General disorders) | 53 (53) — This symptom was assessed as a solicited general AE,
Myalgia (General disorders) | 64 (64) — This symptom was assessed as a solicited general AE.
Arthralgia (General disorders) | 34 (34) — This symptom was assessed as a solicited general AE.
Headache (Nervous system disorders) | 73 (73) — This symptom was assessed as a solicited general AE.
Rash (Skin and subcutaneous tissue disorders) | 74 (74) — This symptom was assessed as a solicited general AE.
Fever (General disorders) | 87 (87) — This symptom was assessed as a solicited general AE.
Bronchitis (Infections and infestations) | 21 (21)
Nasopharyngitis (Infections and infestations) | 31 (31)
Pharyngitis (Infections and infestations) | 13 (13)
Gastroenteritis (Infections and infestations) | 5 (5)
Bronchiolitis (Infections and infestations) | 11 (11)
Otitis media (Infections and infestations) | 6 (6)
Pneumonia (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 6 (6)
Conjunctivitis (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 4 (4)
Acute sinusitis (Infections and infestations) | 2 (2)
Herpangina (Infections and infestations) | 2 (2)
Laryngitis (Infections and infestations) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 8 (8)
Injection site erythema (General disorders) | 9 (9)
Injection site induration (General disorders) | 7 (7)
Injection site pruritus (General disorders) | 7 (7)
Injection site pain (General disorders) | 2 (2)
Injection site warmth (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Colitis (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eating disorder (Psychiatric disorders) | 6 (6)
Irritability (Psychiatric disorders) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Nail injury (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Lymphadentitis (Blood and lymphatic system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Prostatic cyst (Reproductive system and breast disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Bronchitis (Infections and infestations) | 94 (100) — This symptom was assessed as a MAAE.
Nasopharyngitis (Infections and infestations) | 82 (93) — This symptom was assessed as a MAAE.
Pharyngitis (Infections and infestations) | 40 (42) — This symptom was assessed as a MAAE.
Gastroenteritis (Infections and infestations) | 30 (31) — This symptom was assessed as a MAAE.
Bronchiolitis (Infections and infestations) | 28 (29) — This symptom was assessed as a MAAE.
Otitis media (Infections and infestations) | 22 (22) — This symptom was assessed as a MAAE.
Pneumonia (Infections and infestations) | 15 (16) — This symptom was assessed as a MAAE.
Rhinitis (Infections and infestations) | 13 (13) — This symptom was assessed as a MAAE.
Conjunctivitis (Infections and infestations) | 12 (12) — This symptom was assessed as a MAAE.
Tonsillitis (Infections and infestations) | 17 (17) — This symptom was assessed as a MAAE.
Upper respiratory tract infection (Infections and infestations) | 11 (11) — This symptom was assessed as a MAAE.
Influenza (Infections and infestations) | 8 (8) — This symptom was assessed as a MAAE.
Cellulitis (Infections and infestations) | 6 (6) — This symptom was assessed as a MAAE.
Acute sinusitis (Infections and infestations) | 5 (5) — This symptom was assessed as a MAAE.
Impetigo (Infections and infestations) | 5 (5) — This symptom was assessed as a MAAE.
Herpes dermatitis (Infections and infestations) | 4 (4) — This symptom was assessed as a MAAE.
Otitis media acute (Infections and infestations) | 4 (4) — This symptom was assessed as a MAAE.
Hand-foot-and-mouth disease (Infections and infestations) | 3 (3) — This symptom was assessed as a MAAE.
Herpangina (Infections and infestations) | 3 (3) — This symptom was assessed as a MAAE.
Laryngitis (Infections and infestations) | 3 (3) — This symptom was assessed as a MAAE.
Oral candidiasis (Infections and infestations) | 3 (3) — This symptom was assessed as a MAAE.
Viral pharyngitis (Infections and infestations) | 3 (3) — This symptom was assessed as a MAAE.
Cystitis (Infections and infestations) | 2 (2) — This symptom was assessed as a MAAE.
Oral herpes (Infections and infestations) | 2 (2) — This symptom was assessed as a MAAE.
Pharyngitis bacterial (Infections and infestations) | 2 (2) — This symptom was assessed as a MAAE.
Pharyngotonsillitis (Infections and infestations) | 2 (2) — This symptom was assessed as a MAAE.
Tracheitis (Infections and infestations) | 2 (2) — This symptom was assessed as a MAAE.
Bacterial infection (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Croup infectious (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Exanthema subitum (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Gastrointestinal infection (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Hordeolum (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Periodontitis (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Pharyngitis streptococcal (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Sinusitis (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Urinary tract infection (Infections and infestations) | 1 (1) — This symptom was assessed as a MAAE.
Pyrexia (General disorders) | 15 (17) — This symptom was assessed as a MAAE.
Injection site erythema (General disorders) | 1 (1) — This symptom was assessed as a MAAE.
Injection site pruritus (General disorders) | 1 (1) — This symptom was assessed as a MAAE.
Oedema peripheral (General disorders) | 2 (2) — This symptom was assessed as a MAAE.
Chest pain (General disorders) | 1 (1) — This symptom was assessed as a MAAE.
Injection site rash (General disorders) | 1 (1) — This symptom was assessed as a MAAE.
Injection site swelling (General disorders) | 1 (1) — This symptom was assessed as a MAAE.
Enteritis (Gastrointestinal disorders) | 22 (23) — This symptom was assessed as a MAAE.
Diarrhoea (Gastrointestinal disorders) | 7 (7) — This symptom was assessed as a MAAE.
Vomiting (Gastrointestinal disorders) | 8 (8) — This symptom was assessed as a MAAE.
Constipation (Gastrointestinal disorders) | 7 (7) — This symptom was assessed as a MAAE.
Stomatitis (Gastrointestinal disorders) | 7 (7) — This symptom was assessed as a MAAE.
Gastritis (Gastrointestinal disorders) | 6 (6) — This symptom was assessed as a MAAE.
Abdominal pain (Gastrointestinal disorders) | 2 (2) — This symptom was assessed as a MAAE.
Colitis (Gastrointestinal disorders) | 3 (3) — This symptom was assessed as a MAAE.
Chronic gastritis (Gastrointestinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Dental caries (Gastrointestinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Gastritis erosive (Gastrointestinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 20 (20) — This symptom was assessed as a MAAE.
Dermatitis (Skin and subcutaneous tissue disorders) | 11 (11) — This symptom was assessed as a MAAE.
Urticaria (Skin and subcutaneous tissue disorders) | 10 (12) — This symptom was assessed as a MAAE.
Dermatitis contact (Skin and subcutaneous tissue disorders) | 8 (8) — This symptom was assessed as a MAAE.
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) — This symptom was assessed as a MAAE.
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) — This symptom was assessed as a MAAE.
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 18 (18) — This symptom was assessed as a MAAE.
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) — This symptom was assessed as a MAAE.
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — This symptom was assessed as a MAAE.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — This symptom was assessed as a MAAE.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — This symptom was assessed as a MAAE.
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This symptom was assessed as a MAAE.
Eating disorder (Psychiatric disorders) | 3 (3) — This symptom was assessed as a MAAE.
Irritability (Psychiatric disorders) | 1 (1) — This symptom was assessed as a MAAE.
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) — This symptom was assessed as a MAAE.
Contusion (Injury, poisoning and procedural complications) | 2 (2) — This symptom was assessed as a MAAE.
Laceration (Injury, poisoning and procedural complications) | 1 (2) — This symptom was assessed as a MAAE.
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) — This symptom was assessed as a MAAE.
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) — This symptom was assessed as a MAAE.
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) — This symptom was assessed as a MAAE.
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — This symptom was assessed as a MAAE.
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — This symptom was assessed as a MAAE.
Dizziness (Nervous system disorders) | 1 (1) — This symptom was assessed as a MAAE.
Conjunctivitis allergic (Eye disorders) | 1 (1) — This symptom was assessed as a MAAE.
Keratitis (Eye disorders) | 1 (1) — This symptom was assessed as a MAAE.
Anaemia (Blood and lymphatic system disorders) | 1 (1) — This symptom was assessed as a MAAE.
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) — This symptom was assessed as a MAAE.
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) — This symptom was assessed as a MAAE.
Haematuria (Renal and urinary disorders) | 1 (1) — This symptom was assessed as a MAAE.
Renal cyst (Renal and urinary disorders) | 1 (1) — This symptom was assessed as a MAAE.
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) — This symptom was assessed as a MAAE.
Ear pain (Ear and labyrinth disorders) | 1 (1) — This symptom was assessed as a MAAE.
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) — This symptom was assessed as a MAAE.
Prostatic cyst (Reproductive system and breast disorders) | 1 (1) — This symptom was assessed as a MAAE.
Orthostatic hypotension (Vascular disorders) | 1 (1) — This symptom was assessed as a MAAE.
Atopy (Immune system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
sleepiness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2012-06-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT01766206/Prot_000.pdf
  • Statistical Analysis Plan (2013-03-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01766206/SAP_001.pdf